CLINICAL TRIAL: NCT02840630
Title: Effect of FISH Intake on MEtabolic Health in a Diabetic South Asian popuLation (FISH MEAL)
Acronym: FISHMEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT10087-10
Record Dates: First submitted 2016-06-14; First posted 2016-07-21 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: n3 LC-PUFA; Type 2 Diabetes Mellitus; South Asian; HbA1c; Omega 3 status
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-diabetic group (No Intervention): Non-diabetic volunteers will be recruited for baseline data. They will only be required to provide dried blood samples (DBS) samples and information at week 0. They have to collect finger prick DBS, weigh themselves and fill in food frequency questionnaire only at one time point.
- Diabetic control intervention group (No Intervention): The diabetic control group will provide finger prick DBS at week 0, 8 and 16, fill in food frequency questionnaire at week 0 and 16 and weekly weighing from week 0 until 16. This group will not be receiving tinned mackerel and will be asked to continue with their habitual diet and lifestyle.
- Diabetic fish intervention group (Active Comparator): This intervention group will receive two 125 g portion of tinned mackerel fish (containing 7.8 g n-3 LCPUFA) per week from week 0 until 16 and a mackerel recipe book each. They will be required to provide finger prick DBS at week 0, 8 and 16, fill in food frequency questionnaire at week 0 and 16 and weekly weighing from week 0 until 16.
  Interventions: Other: Tinned mackerel fish

INTERVENTIONS:
Other: Tinned mackerel fish — Diabetic fish intervention group will be given two tinned mackerels per week from week 0 until week 16.
  Other Names: Tesco tinned mackerel fish
  Arms: Diabetic fish intervention group

SUMMARY:
The investigators will recruit non-diabetic volunteers (n=30) and diabetic volunteers controlled by diet and lifestyle (n=300). The non-diabetic volunteers will be in the non-diabetic group while the diabetic volunteers will be randomised to a diabetic control intervention group or a diabetic fish intervention group. Baseline data will be collected from all three groups but only diabetic control intervention group and diabetic fish intervention group will go through the 16-week study. This will allow the investigators to compare the metabolic health across South Asian population in people with and without diabetes.

The recommended intake of EPA and DHA daily is ~450 mg per day for cardiovascular health, or approximately 3 g per week. Over the course of 16 weeks, subjects in the diabetic control intervention group will continue with their habitual diet, while subjects in the diabetic fish intervention group will receive two 125 g portion of tinned mackerel (containing 7.8 g n-3 LCPUFA26) every week, to replace a portion of red meat or poultry. Previous n-3 LCPUFA intervention study among South Asian people in the United Kingdom was able to reverse lipid abnormalities with supplementation of 2.5 g of EPA and DHA per day for 12 weeks. However, the same study also shows that their daily consumption of EPA and DHA is only 68±99 and 112±171 mg respectively. Therefore, only 1.1 g n-3 LCPUFA per day is given in this study to increase compliance.

Recipe recommendations using mackerel will be provided. Non-diabetic volunteers will be recruited only to obtain baseline data in order to compare their metabolic profile with that of the diabetic volunteers. This will allow us to investigate the link between omega 3 status and glycaemic control in a South Asian population.

Fish is chosen as an intervention as opposed to EPA and DHA supplements in order to capture the benefits of eating fish as an important source of not only n-3 LCPUFA, but also other key nutrients such as vitamin D, selenium and iodine.

DETAILED DESCRIPTION:
During the study period, participants will be asked to maintain their routine dietary and social habits to avoid changes in body weight. In addition volunteers will be asked to record their weights first thing in the morning on the same set of scales every week. Any changes can be documented in a food frequency questionnaire. Volunteers without diabetes will be recruited for baseline data and will not be involved in the 16-week intervention study. Diabetic volunteers will be randomized by BioSS in batches of ~20 people into the diabetic control or the diabetic fish intervention group that will be matched for gender, age and BMI. The diabetic control group will be asked to continue with their routine dietary habits while the diabetic fish intervention group will be asked to substitute poultry or red meat with 2 tins of mackerels each week. Study kits will be posted two weeks before the study initiates to consenting volunteers.

All volunteers will be asked to provide finger prick blood spots on filter paper at week 0, while subjects allocated to diabetic control and diabetic fish intervention groups will be asked to provide blood spots again at week 8 and 16. A dried blood spot (DBS) sampling kit containing two Whatman 903 filter papers, two lancets, alcohol pads, bandaids, guidelines on spotting blood on filter paper, prepaid envelope, FFQ, tinned mackerel and a fish recipe book. Every volunteer will be asked to prick the inside tip of a non-dominant finger and gently spot a total of ten circles in the filter papers. A volunteer might experience slight discomfort when the lancet goes into the finger. The volunteers will then allow the filter paper to dry for about an hour before closing the flap over the filter paper. All information and tools to help with obtaining the dried blood spots, as well as guidelines on how to spot blood on filter paper will be included with the DBS kit. Volunteers are required to spot 2 filter papers at one collection point and post them in a pre-paid envelope complete with a return address.

The DBS samples will be analyzed for omega 3 index, glycated hemoglobin (HbA1c), triglycerides, Vitamin D status, genetic (TCF7L2 7903146) and epigenetic marker (FADS 174546) of lipid and glucose control.

ELIGIBILITY:
Non-diabetic group:

Inclusion Criteria

* Of South Asian origin (defined by country of birth, last name and self-report ethnicity)
* Men and women between the age of 25 and 65;
* Body mass index (BMI) of ≥23 kg/m2 according to WHO classification for Asian population;
* Ability to speak, read and understand the English language.

Exclusion criteria

* Use of tobacco;
* Use of insulin or oral hypoglycaemic agents;
* Use of medications that are known to affect lipid metabolism,
* Haemophiliacs,
* Use of medications that are known to generally alter the haemostatic system;
* Diagnosis of diabetes;
* Diagnosis of hypertension, renal, hepatic, haematological disease or coronary heart disease;
* Have previously donated blood for transfusion purposes within the last month;
* Inability to understand participant information sheet.

Diabetic control intervention and diabetic fish intervention group:

Inclusion Criteria

* Of South Asian origin (defined by country of birth, last name and self-report ethnicity)
* Men and women between the age of 25 and 65;
* Body mass index (BMI) of ≥23 kg/m2 according to WHO classification for Asian population;
* Diagnosed with diabetes only controlled by diet and lifestyle;
* Ability to speak, read and understand the English language.

Exclusion criteria

* Use of tobacco;
* Use of insulin or oral hypoglycemic agents;
* Use of medications that are known to affect lipid metabolism;
* Haemophiliacs;
* Use of medications that are known to generally alter the hemostatic system;
* Diagnosis of hypertension, renal, hepatic, haematological disease or coronary heart disease;
* Have previously donated blood for transfusion purposes within the last month;
* Inability to understand participant information sheet.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) | week 0 and 16
  HbA1c will be analysed from DBS samples at week 0 and 16.

SECONDARY OUTCOMES:
Change in Omega 3 Index | week 0, 16
  Omega 3 Index will be analysed from DBS samples at week 0, and 16.
Change in Triglycerides | week 0, and 16
  Triglycerides will be analysed from DBS samples at week 0 and 16.
Change in Vitamin D | week 0, 16
  Vitamin D will be analysed from DBS samples at week 0 and 16.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje De Roos, BSc, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No